CLINICAL TRIAL: NCT06213428
Title: Investigating the Effects of Probiotics on Synaptic Plasticity in the Follicular and Luteal Phases of the Menstrual Cycle
Brief Title: Effects of Probiotics on Synaptic Plasticity During the Menstrual Cycle
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Aimee Nelson, Dr., McMaster University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16602
Record Dates: First submitted 2023-12-26; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Women's Health; Brain Plasticity
Keywords: Probiotic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: all investigators and participants will be masked to which condition they receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active: Probiotic (Active Comparator): Progressive Perfect Probiotic 120 Billion CFU containing the following strains will be used:
  Lactobacillus plantarum, Lactobacillus rhamnosus, Lactobacillus acidophilus, Bifidobacterium animalis subsp.lactis, Bifidobacterium breve, Lactobacillus paracasei, Lactobacillus casei, Lactobacillus gasseri, Lactobacillus reuteri, Bifidobacterium bifidum, Bifidobacterium longum subsp. Longum.
  Participants will be required to take one capsule a day, for 28 days.
  Interventions: Biological: Progressive Perfect Probiotic
- Placebo Probiotic (Placebo Comparator): A placebo that is identical in capsule size and colour to the active probiotic capsule will be used. This will ensure participants and experimenters are masked during each intervention period. Participants will be required to take one capsule a day for 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Progressive Perfect Probiotic — Participants will be administered an active probiotic for 28 days. Participants will be blinded as to what intervention they are experiencing.
  Arms: Active: Probiotic
Other: Placebo — Participants will be administered a placebo for 28 days. Participants will be blinded as to what intervention they are experiencing.
  Arms: Placebo Probiotic

SUMMARY:
Modulation of our gut microbiota through probiotics, can improve our emotional state, decrease pain sensitivity, improve cognitive processes, increase neurotransmitter levels and alter functional connectivity. In addition, probiotics regulate estrogen levels. Estrogen levels have been recognized to influence the gut microbiota, impact neural activity, memory, and cognition.

This study aims 1) to determine whether probiotics can increase the propensity for synaptic plasticity in females and 2) to determine if there are differences in the propensity for plasticity depending on the phase of the menstrual cycle.

DETAILED DESCRIPTION:
The human gastrointestinal (GI) tract is comprised of trillions of bacterial strains. Recent work has focused on investigating the influence of the gut microbiota on the processing and function of our brain; this is known as the 'gut-brain axis'. Our gut microbiota can be altered through diet, antibiotics, prebiotics and probiotics (Hemarajata et al., 2013). Probiotics are live microorganisms, which when delivered in adequate amounts, can offer beneficial health outcomes to the host (Hill et al., 2014). Modulation of our gut microbiota through probiotics, can improve our emotional state (Bagga et al., 2018; Messaoudi et al., 2011; Tillisch et al., 2013), decrease pain sensitivity (Weizman et al., 2016), improve cognitive processes (Chung et al., 2014; Kim et al., 2020), increase neurotransmitter levels (Mittal et al., 2017) and alter functional connectivity (Rode et al., 2022; Bagga et al., 2019). In addition, probiotics regulate estrogen levels (Guo et al., 2016; Urbaniak et al., 2016).

Estrogen levels have been recognized to influence the gut microbiota. The gut produces β-glucuronidases which is the enzyme required to breakdown conjugated estrogen into its active form (Dabek et al., 2008; Ervin et al., 2019). Low β-glucuronidases production occur in the presence of diminished bacterial diversity levels in the gut. The consequence of the low β-glucuronidases is a reduction in active forms of estrogen (Siddiqui et al., 2022; Pugh et al., 2021; Kwa et al., 2016, Baker et al., 2017). Further, gastrointestinal symptoms increase during menstruation (Pugh et al., 2021). Last, irritable bowel syndrome is more prevalent in females, indicating a possible role of sex hormones in relation to the gut microbiome (Pugh et al., 2021).

Estrogen has been found to impact neural activity, memory, and cognition (Inghilleri et al., 2004; Luine 2014). EEG brain activity was collected from women in their follicular and luteal phase (Brotzner et al., 2014). When estrogen levels were highest, individual alpha frequency oscillations (IAF) were lowest (Brotzner et al., 2014), the latter is associated with reduced cognition and working memory (Li et al., 2023). In addition, estrogen was found to reduce the firing threshold in some neurons which can promote excitability in the cortex (Gregory et al., 2019). Conversely, high progesterone levels are known to increase GABA activity which reduces neural activity (Guennoun et al., 2015). Furthermore, a 5Hz repetitive transcranial magnetic stimulation (rTMS) protocol was delivered over the motor cortex during the early and late follicular phase (Inghilleri et al., 2004). Corticospinal activity was increased when estradiol levels were highest (Inghilleri et al., 2004) showing the association between estradiol and synaptic plasticity.

Collectively, the literature suggests that women may have a reduced capacity for synaptic plasticity during the luteal phase when estradiol levels are low. Introducing a probiotic will increase β-glucuronidases which leads to greater availability of circulating estrogen which should promote synaptic plasticity. It is hypothesized that increases in synaptic plasticity will occur in the follicular and luteal phase in the presence of probiotics. This study aims 1) to determine whether probiotics can increase the propensity for synaptic plasticity in females and 2) to determine if there are differences in the propensity for plasticity depending on the phase of the menstrual cycle.

Methods:

Participants will be randomized into Group A or Group B. Twenty participants will be in Group A and 20 participants will be in group B. If randomized to Group A, all visits will be conducted between day 6-9 (mid-follicular phase) when estradiol levels are highest. If randomized to Group B, all visits will be conducted during day 19-23 (mid-luteal phase) when progesterone levels are highest. This will be a randomized, crossover, double-masked study whereby participants will receive both real probiotic and placebo probiotic for 28 days. Assessments will be acquired during four visits (Before and after each intervention, separated by a 28 day washout). The McMaster University Medical Centre (MUMC) pharmacy will be responsible for the preparation of the blinded probiotic kits and randomization schedule. The probiotic used will be a commercially available product called Progressive Perfect Probiotic (https://www.progressivenutritional.com/products/perfect-probiotic-120-billion).

The following dependent measures will be used: Active motor threshold, Resting motor threshold, short interval intracortical inhibition, motor evoked potentials.

These measures will be taken before and after a synaptic plasticity inducing protocol

To assess synaptic plasticity, repetitive TMS will be performed using a 70mm inner diameter figure-of-eight coil with a Magstim Super Rapid2 Plus Stimulator (Magstim, Whitland, UK). Biphasic magnetic pulses will be delivered over the primary motor area of the dominant hemisphere to find the optimal position for eliciting a MEP in the contralateral APB muscle. Intermittent theta burst stimulation (iTBS) protocol will be delivered using biphasic pulses in burst of three pulses delivered in 6Hz trains that will last 2s, this will be followed by 8s with no pulse delivered. iTBS will be repeated for a total of 612 pulses at 80% of AMT (Fassett et al., 2017).

ELIGIBILITY:
Inclusion Criteria:

* right handed, females between 18-35 years old with a regular menstrual cycle (approximately 26-30 days)

Exclusion Criteria:

* contradictions to TMS
* contradictions to probiotic
* Females who use hormone altering devices (i.e. oral contraceptives)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change Motor Evoked Potentials (MEPs) | Immediately before intervention, immediately following 4 week intervention
  Change in MEPs using TMS

SECONDARY OUTCOMES:
Short Interval intracortical inhibition (SICI) | Immediately before intervention, immediately following 4 week intervention
  Changes in SICI Using TMS

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Unviersity, Hamilton, Ontario, Canada